CLINICAL TRIAL: NCT06951282
Title: Impact of Selenium on Methotrexate Induced Spermatotoxicity; A Comparative Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD70/2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Methotrexate Spermatotoxicity
MeSH Terms: interventions — Selenium; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No selenium or methotrexate group (No Intervention): no selenium or methotrexate were given
- Selenium group (Active Comparator): 200 microgram selenium was given daily for 3 months
  Interventions: Dietary Supplement: Selenium
- Methotrexate group (Active Comparator): 0.4 mg/kg/week subcutaneous methotrexate was given for 3 months
  Interventions: Drug: Methotrexate
- Selenium and methotrexate group (Active Comparator): 200 microgram selenium was given daily for 3 months along with 0.4 mg/kg/week subcutaneous methotrexate for 3 months
  Interventions: Dietary Supplement: Selenium; Drug: Methotrexate

INTERVENTIONS:
Dietary Supplement: Selenium — 200 microgram selenium was given daily for 3 months
  Arms: Selenium and methotrexate group; Selenium group
Drug: Methotrexate — 0.4 mg/kg/week sub cutaneous methotrexate for 3 months
  Arms: Methotrexate group; Selenium and methotrexate group

SUMMARY:
The aim of this study is to assess the potential protective role of selenium on semen parameters and its effect on seminal glutathione peroxidase level in patients on MTX therapy

DETAILED DESCRIPTION:
The aim of this study is to assess the potential protective role of selenium on semen parameters and its effect on seminal glutathione peroxidase level in patients on MTX therapy. informed consent was obtained from each patient after explanation of the purpose of the study. All patients were subjected to history taking and general and local examination. Baseline semen analysis and seminal glutathione peroxidase (GPX) were done for all patients and then they were divided into four groups each has 10 patients.

The no Se or MTX group was not eligible for neither Se nor MTX intake. The Se group started Se intake in a daily dose of 200 µg according to the United States National Academy of Sciences for 3 months.

Patients of both MTX groups (MTX group & MTX and Se group) were chosen from psoriatic patients already planned to start MTX treatment with subcutaneous dose of 0.3-0.4 mg/kg/week.

The MTX and Se group started Se intake in a daily dose of 200 µg according to the United States National Academy of Sciences for 3 months.

After 3 months, semen analysis and seminal GPX level were repeated.

ELIGIBILITY:
Inclusion Criteria:

* adult males from 18-60 years old for the 2 methotrexate (MTX) study groups, the males included were chosen from patients already planned to start MTX treatment for psoriasis

Exclusion Criteria:

* History of drug intake that can affect semen parameters i.e., cytotoxic drugs, anti-androgens, sulfasalazine, gonadal hormones, nitrofurans or salicylic acid within previous three months.
* History of smoking within the last three months.
* Chronic disorders such as diabetes mellitus, hypertension, obesity, chronic liver or renal disease.
* Organic diseases that can affect fertility i.e., varicocele, testicular tumor or undescended testis.
* Genitourinary diseases.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Glutathione peroxidase level | from enrollment to 3 months
  Seminal glutathione peroxidase level was measured in the four studied groups at baseline and after 3 month duration
semen volume | from enrollment to 3 months
  Semen volume in (ml) was measured in all patients of the 4 studied groups at baseline and after 3 months
Sperm count / ejaculate | from enrollment to 3 months
  Sperm count / ejaculate in (million) was measured in all patients of the 4 studied groups at baseline and after 3 months
Sperm concentration / ml | from enrollment to 3 months
  Sperm concentration / ml in (million) was measured in all patients of the 4 studied groups at baseline and after 3 months
Sperm motility | from enrollment to 3 months
  percentage of sperm progressive, non progressive and total motility were measured in all patients of the 4 studied groups at baseline and after 3 months
Sperm morphology | from enrollment to 3 months
  percentage of sperms with normal morphology was measured in all patients of the 4 studied groups at baseline and after 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt